CLINICAL TRIAL: NCT04166773
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study Comparing the Efficacy and Safety of Tirzepatide Versus Placebo in Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Nonalcoholic Steatohepatitis (NASH)
Acronym: SYNERGY-NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17361; I8F-MC-GPHR (Other: Eli Lilly and Company); 2019-001550-26 (EudraCT Number)
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo administered SC once a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the study drug, tirzepatide administered once weekly, is safe and effective as a treatment for Nonalcoholic Steatohepatitis (NASH).

ELIGIBILITY:
* Participants must have a body mass index (BMI) ≥27 kilograms per square meter (kg/m²) and ≤50 kg/m² with stable body weight for at least 3 months
* Participants with or without type 2 diabetes mellitus (T2DM)

  * If with T2DM, hemoglobin A1c (HbA1c) ≤9.5%
* Participants must be willing to undergo baseline and endpoint liver biopsies
* Participants must have histologic diagnosis of NASH with stage 2 or 3 fibrosis by liver biopsy
* Participants must not have known or suspected alcohol abuse (>14 units/week for women and >21 units/week for men) or active substance abuse
* Participants must not have evidence of cirrhosis or other forms of liver disease
* Participants must not have heart attack, stroke, or hospitalization for congestive heart failure in the past 6 months
* Participants must not have active cancer within the last 5 years
* Participants must not have uncontrolled high blood pressure
* Participants must not have renal impairment with estimated glomerular filtration rate (eGFR) <30 milliters/minute/1.73m²; for participants on metformin, eGFR <45 mL/min/1.73m²
* Participants must not have a diagnosis of type 1 diabetes
* Participants must not have a history of pancreatitis (acute or chronic)
* Participants must not have calcitonin ≥35 nanograms per liter
* Participant must not have family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (family is defined as a first degree relative)
* Female participants must not be pregnant, breast-feeding, or intend to become pregnant or of childbearing potential and not using adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (112):
- United States (47):
  - University of Alabama-The Kirklin Clinic, Birmingham, Alabama
  - Synexus Clinical Research US, Inc., Chandler, Arizona
  - Fresno Clinical Research Center, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Diabetes Medical Center of California, Northridge, California
  - Velocity Clinical Research, Panorama City, Panorama City, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - IHS Health Research, Kissimmee, Florida
  - Accel Research Sites - Maitland Clinical Research Unit, Maitland, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - The Center for Digestive Health, Orlando, Florida
  - Synexus Clinical Research US, Inc., Orlando, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Synexus Clinical Research, Chicago, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - The National Diabetes & Obesity Research Institute, Biloxi, Mississippi
  - Southern Therapy and Advanced Research (STAR) LLC, Jackson, Mississippi
  - Buffalo Clinical and Translational Research Center, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Radiant Research - Dallas North, Dallas, Texas
  - Liver Center of Texas, PLLC, Dallas, Texas
  - Texoma Medical Center, Denison, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - National Clinical Research, Inc, Richmond, Virginia
  - Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
  - Harborview Medical Center/University of Washington, Seattle, Washington
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerpen
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Delta vzw, Roeselare, West-Vlaanderen
- France (7):
  - CHU Bordeaux Haut-Leveque, Pessac, Aquitaine
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges, Haute-Vienne
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine-et-Loire
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Pitie Salpetriere University Hospital, Paris
  - Hôpital Saint Antoine, Paris
- Israel (6):
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Galilee Medical Center, Nahariya, Northern District
  - Carmel Hospital, Haifa
- Italy (5):
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Di Foggia, Foggia
  - Ospedale Santa Maria Goretti, Latina
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Japan (16):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - JCHO Hokkaido Hospital, Sapporo, Hokkaido
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - JADECOM Nara City Hospital, Nara, Nara
  - Hirakata kohsai Hospital, Higashi-cho, Hirakata-city, Osaka
  - Osaka Saiseikai Suita hospital, Suita, Osaka
  - Shimane University Hospital, Izumo, Shimane
  - Tokyo Medical And Dental University Medical Hospital, Bunkyō, Tokyo
  - Fukuiken Saiseikai Hospital, Fukui
  - Gifu Municipal Hospital, Gifu
  - Kumamoto Shinto General Hospital, Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Saga University Hospital, Saga
  - Yamagata University Hospital, Yamagata
- Mexico (4):
  - Phylasis Clinicas Research, Cuautitlan Izcalli, Mexico City
  - Grupo Medico Camino Sc, Mexico City, Mexico City
  - Christus Muguerza Hospital Sur, Monterrey, Nuevo León
  - Centro de Investigación y Gastroenterología, Cuauhtémoc
- Poland (2):
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - Synexus Polska Oddział w Lodzi, Lodz, Łódź Voivodeship
- Spain (7):
  - Clínica Juaneda, Palma de Mallorca, Balears [Baleares]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Instituto de Ciencias Médicas, Alicante
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (13):
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Synexus North East Clinical Research Centre, Hexham, England
  - Royal London Hospital, London, England
  - St. George's Hospital, London, England
  - Synexus Clinical Research Centre - Lancashire, Chorley, Lancashire
  - King's College Hospital, London, London, City of
  - Queen's Medical Centre, Nottingham University Hospitals, Nottingham, Nottinghamshire
  - John Radcliffe Hospital, Headington, Oxford
  - Synexus North Teesside Clinical Research Centre, Stockton-on-Tees, Stockton-on-Tees
  - Imperial College London - St Mary's Hospital, London, Westminster
  - Synexus Midlands Clinical Research Centre, Birmingham
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Synexus Manchester Clinical Research Centre, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Loomba R, Hartman ML, Lawitz EJ, Vuppalanchi R, Boursier J, Bugianesi E, Yoneda M, Behling C, Cummings OW, Tang Y, Brouwers B, Robins DA, Nikooie A, Bunck MC, Haupt A, Sanyal AJ; SYNERGY-NASH Investigators. Tirzepatide for Metabolic Dysfunction-Associated Steatohepatitis with Liver Fibrosis. N Engl J Med. 2024 Jul 25;391(4):299-310. doi: 10.1056/NEJMoa2401943. Epub 2024 Jun 8. PMID 38856224
- See also: A Study of Tirzepatide (LY3298176) in Participants With Nonalcoholic Steatohepatitis (NASH) — https://trials.lillytrialguide.com/en-US/trial/3lQTuBFU3GBu9vi4SAlDDp

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Milligram (mg) Tirzepatide: Participants received 5 mg tirzepatide administered subcutaneously (SC) once a week (QW) for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks, then 5 mg tirzepatide SC QW from weeks 5-52].
- 10 mg Tirzepatide: Participants received 10 mg tirzepatide administered SC QW for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks, then dose escalated to 5 mg, 7.5 mg, and 10 mg every 4 weeks until target dose (10 mg) was reached].
- 15 mg Tirzepatide: Participants received 15 mg tirzepatide administered SC QW for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks, then dose escalated to 5 mg, 7.5 mg, 10 mg, 12.5 mg, and 15 mg every 4 weeks until target dose (15 mg) was reached].
- Placebo: Participants received placebo administered SC QW for 52 weeks.
Period: Overall Study
Arm/Group | 5 Milligram (mg) Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 47 | 47 | 48 | 48
Received at Least One Dose of Study Drug | 47 | 47 | 48 | 48
Completed | 40 | 44 | 43 | 38
Not Completed | 7 | 3 | 5 | 10
Not completed — Adverse Event | 2 | 0 | 2 | 1
Not completed — Lost to Follow-up | 4 | 2 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC QW for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks, then 5 mg tirzepatide SC QW from weeks 5-52].
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 47 | 47 | 48 | 48 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.00 (11.62) | 54.30 (12.08) | 54.90 (10.02) | 53.50 (11.60) | 54.40 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 29 | 27 | 109
  Male | 20 | 21 | 19 | 21 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 17 | 18 | 69
  Not Hispanic or Latino | 21 | 25 | 27 | 24 | 97
  Unknown or Not Reported | 7 | 7 | 4 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 0 | 3
  Asian | 5 | 6 | 6 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 41 | 39 | 41 | 43 | 164
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 1 | 0 | 1
  France | 7 | 7 | 2 | 6 | 22
  Israel | 3 | 2 | 0 | 0 | 5
  Italy | 1 | 0 | 2 | 3 | 6
  Japan | 4 | 4 | 4 | 4 | 16
  Mexico | 1 | 3 | 3 | 3 | 10
  Poland | 1 | 0 | 0 | 0 | 1
  Spain | 1 | 0 | 6 | 1 | 8
  United Kingdom | 1 | 5 | 4 | 4 | 14
  United States | 28 | 26 | 26 | 27 | 107

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Absence of Nonalcoholic Steatohepatitis (NASH) With no Worsening of Fibrosis on Liver Histology
Description: NASH resolution is defined as the absence of fatty liver disease or simple steatosis without steatohepatitis; the absence of hepatocellular ballooning (nonalcoholic fatty liver disease (NAFLD) Activity Score (NAS) 0 for ballooning); with or without mild lobular inflammation (NAS 0 or 1 for inflammation); and any value for steatosis. No worsening of fibrosis is defined as no increase in fibrosis stage from baseline to Week 52.
Time Frame: Week 52
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline values and had evaluable data for this outcome prior to treatment discontinuation.
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 39 | 41 | 40 | 35
Percentage of participants | 51.84 | 63.13 | 73.92 | 12.62
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.45, 95% CI 2-sided [2.27 to 24.44] — Odds ratio, Confidence Interval (CI), and p-value for endpoint measures are from logistic regression model with baseline diabetes status, region, treatment as factors
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.86, 95% CI 2-sided [3.59 to 39.11] — Odds ratio, CI, and p-value for endpoint measures are from logistic regression model with baseline diabetes status, region, treatment as factors
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 19.63, 95% CI 2-sided [5.73 to 67.25] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With ≥1 Point Decrease in Fibrosis Stage With No Worsening of NASH on Liver Histology
Description: NAS was derived as the unweighted sum of steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocellular ballooning (0 to 2) scores. The NAS ranges from 0-8 with the higher score indicating more aggressive disease. Evaluation of fibrosis stage was based on the nonalcoholic steatohepatitis clinical research network (NASH CRN) fibrosis staging system, which was scaled from 0 to 4 stages where, 0=None to 4=Cirrhosis. Participants were evaluated with the NASH CRN scoring system with ≥1-point reduction without worsening of NASH (defined as no increase in the NAS score).
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC QW for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks then 5 mg tirzepatide SC QW from week 5-52].
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 39 | 41 | 40 | 35
Percentage of participants | 59.21 | 53.35 | 54.3 | 32.51
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.025, Regression, Logistic; Odds Ratio (OR) = 3.01, 95% CI 2-sided [1.15 to 7.90] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.074, Regression, Logistic; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.92 to 6.13] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.063, Regression, Logistic; Odds Ratio (OR) = 2.47, 95% CI 2-sided [0.95 to 6.40] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants With ≥1 Point Increase in Fibrosis Stage on Liver Histology
Description: Participants were evaluated with the NASH CRN scoring system with ≥1 stage increase in fibrosis.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 39 | 41 | 40 | 35
Percentage of participants | 12.04 | 9.81 | 5.53 | 13.03
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.893, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.25 to 3.40] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.647, Regression, Logistic; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.18 to 2.87] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p = 0.246, Regression, Logistic; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.08 to 1.91] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants That Achieve a ≥2 Point Decrease in NAFLD (Non-alcoholic Fatty Liver Disease) Activity Score (NAS) on Liver Histology, With ≥1 Point Reduction in at Least 2 NAS Components
Description: Hepatic histological improvement in NAS was defined as a decrease (improvement) in NAS by ≥ 2 with at least a 1-point reduction in at least 2 NAS components (lobular inflammation, hepatocellular ballooning or steatosis). The NAS was derived as the unweighted sum of steatosis (0 to 3), lobular inflammation (0 to 3), and hepatocellular ballooning (0 to 2) scores. The NAS ranges from 0-8, with the higher score indicating more aggressive disease.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 39 | 41 | 40 | 35
Percentage of participants | 81.02 | 86.55 | 88.77 | 38.09
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.94, 95% CI 2-sided [2.41 to 20.00] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.46, 95% CI 2-sided [3.36 to 32.61] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.85, 95% CI 2-sided [3.87 to 42.65] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Mean Absolute Change From Baseline in Liver Fat Content by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF)
Description: MRI-PDFF is an established method that enables quantification of fat content in the liver. The value of whole liver fat as assessed by MRI-PDFF is expressed in percentage (%) and ranges from 0 to 100% with higher values representing higher liver fat level. Least square (LS) mean was calculated using mixed model repeated measures (MMRM) model for post-baseline measures: Variable = Baseline + Diabetes Flag (DIABFL) + REGION1 + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: absolute percentage of liver fat
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 28 | 33 | 32 | 27
absolute percentage of liver fat | -10.12 (1.165) | -10.15 (1.071) | -11.34 (1.107) | -1.31 (1.142)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -8.81, 95% CI 2-sided [-12.04 to -5.58], Standard Error of Mean 1.632
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -8.83, 95% CI 2-sided [-11.93 to -5.73], Standard Error of Mean 1.566
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.02, 95% CI 2-sided [-13.17 to -6.87], Standard Error of Mean 1.591

6. Secondary Outcome: Mean Change From Baseline in Body Weight
Description: Change in body weight at the end of 52 weeks measured in kilogram (kg) using a calibrated scale. LS mean was calculated using MMRM model for post-baseline measures: Variable = Baseline + DIABFL + REGION1 + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC QW for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks, then 5 mg tirzepatide SC QW from week 5-52].
- 10 mg Tirzepatide: Participants received 10 mg tirzepatide administered SC QW for 52 weeks [initially 2.5 mg tirzepatide SC QW for 4 weeks, then dose escalated to 5 mg, 7.5 mg and 10 mg every 4 weeks until target dose (10 mg) was reached].
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 40 | 42 | 42 | 37
Kilogram (kg) | -11.46 (1.404) | -14.22 (1.380) | -17.88 (1.376) | -1.04 (1.392)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.42, 95% CI 2-sided [-14.32 to -6.52], Standard Error of Mean 1.976
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -13.19, 95% CI 2-sided [-17.05 to -9.32], Standard Error of Mean 1.960
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -16.84, 95% CI 2-sided [-20.71 to -12.98], Standard Error of Mean 1.957

ADVERSE EVENTS:
Time Frame: Baseline Up to Week 56
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at Risk adjusted accordingly
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 5/47 | 4/47 | 0/48 | 3/48
Other Adverse Events (participants affected / at risk) | 43/47 | 43/47 | 44/48 | 40/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=47) | 10 mg Tirzepatide (N=47) | 15 mg Tirzepatide (N=48) | Placebo (N=48)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/27 (0) | 0/26 (0) | 0/29 (0) | 1/27 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0/27 (0) | 0/26 (0) | 0/29 (0) | 1/27 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=47) | 10 mg Tirzepatide (N=47) | 15 mg Tirzepatide (N=48) | Placebo (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (8) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (12) | 3 (4) | 4 (7) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 6 (10) | 2 (2) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic angioectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (12) | 9 (12) | 7 (8) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 17 (40) | 13 (20) | 11 (14)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 8 (11) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (4) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (5) | 4 (5) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (69) | 16 (33) | 21 (26) | 6 (7)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (5) | 7 (14) | 1 (1)
Asthenia (General disorders) | 3 (3) | 4 (6) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Energy increased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 4 (5) | 5 (5) | 3 (4)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (5) | 1 (2) | 2 (10) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0/27 (0) | 1/26 (1) | 0/29 (0) | 0/27 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 5 (6) | 6 (6) | 9 (9) | 4 (5)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (4) | 2 (2) | 4 (4)
Viral rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0/27 (0) | 0/26 (0) | 1/29 (1) | 0/27 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/27 (0) | 1/26 (1) | 0/29 (0) | 0/27 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biopsy liver (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (3) | 1 (1) | 3 (4) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 3 (3) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 10 (12) | 11 (12) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/27 (0) | 0/26 (0) | 0/29 (0) | 1/27 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 6 (7) | 4 (4) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 6 (7) | 3 (4) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (17) | 0 (0) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/20 (0) | 0/21 (0) | 0/19 (0) | 1/21 (1)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/27 (0) | 0/26 (0) | 1/29 (1) | 0/27 (0)
Testicular pain (Reproductive system and breast disorders) | 0/20 (0) | 0/21 (0) | 0/19 (0) | 1/21 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/27 (0) | 0/26 (0) | 1/29 (1) | 0/27 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0/27 (0) | 0/26 (0) | 0/29 (0) | 1/27 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 3 (5) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Koilonychia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cyst removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid cyst removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nail operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon sheath incision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polypectomy (Surgical and medical procedures) | 0/27 (0) | 0/26 (0) | 1/29 (1) | 0/27 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT04166773/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT04166773/SAP_001.pdf